CLINICAL TRIAL: NCT04718051
Title: S.P.PRO LIVER POWDER is Used to Improve Liver and Metabolic Indexes in People With Non-alcoholic Fatty Liver Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Sheng Pu Pharmaceutics Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202007032
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shen Pu Yang Gan Wan (Experimental): Traditional Chinese Medicine
  Interventions: Drug: Shen Pu Yang Gan Wan
- Placebo Comparator (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Shen Pu Yang Gan Wan — Shen Pu Yang Gan Wan is Traditional Chinese Medicine; in addition, it has a high dose.
  Arms: Shen Pu Yang Gan Wan
Drug: Placebo — Shen Pu Yang Gan Wan is Traditional Chinese Medicine; however, it has a very low dose.
  Arms: Placebo Comparator

SUMMARY:
With the Westernization of the diet and insufficient exercise, Taiwan's population of obesity, diabetes, and hyperlipidemia has increased in recent years, and the prevalence of the non-alcoholic fatty liver disease has gradually increased. Although weight loss, dietary adjustments, and certain drug treatments can delay the deterioration of the disease; however, weight loss and dietary adjustment are not easy.

DETAILED DESCRIPTION:
With the Westernization of the diet and insufficient exercise, Taiwan's population of obesity, diabetes, and hyperlipidemia has increased in recent years, and the prevalence of the non-alcoholic fatty liver disease has gradually increased. Although weight loss, dietary adjustments, and certain drug treatments can delay the deterioration of the disease; however, weight loss and dietary adjustment are not easy. Moreover, drugs also have side effects, and there is currently no convenient and effective treatment for people who have non-alcoholic fatty liver disease. The purpose of this trial is that investigating and evaluating the effects on fatty liver, liver fiber, and metabolic indexes after subjects using Shen Pu Yang Gan Wan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fatty liver diagnosed by abdominal ultrasound or hepatic fibrometer within half a year's data
* Subjects with the non-alcoholic fatty liver disease
* The severity of fatty liver should be at least 3 points by taking an abdominal ultrasound

Exclusion Criteria:

* Female patients are pregnant or breastfeeding.
* Patients with viral hepatitis.
* Long-term drinkers.
* Those who use slimming products and vitamin E.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in AST index | 36 weeks
  Measure the changes in the index which is AST relate to Liver inflammation
Change in ACT index | 36 weeks
  Measure the changes in the index which is ACT relate to Liver inflammation
Change in HbA1c | 36 weeks
  Measure the changes in the index which is HbA1c relate to Liver inflammation
Fibroscan | 36 weeks
  Measure the changes in the index which is Liver Fibrosis

SECONDARY OUTCOMES:
Measuring Body Mass Index | 36 weeks
  Measuring Body Mass Index (BMI). Measure the changes in index which is Metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shun Wu, Study Director — Taipei Municipal Wanfang Hospital
Locations (1):
- Wanfang Hospital, Taipei, Wenshan District, Taiwan

REFERENCES:
- [Background] Yang MD, Chiang YM, Higashiyama R, Asahina K, Mann DA, Mann J, Wang CC, Tsukamoto H. Rosmarinic acid and baicalin epigenetically derepress peroxisomal proliferator-activated receptor gamma in hepatic stellate cells for their antifibrotic effect. Hepatology. 2012 Apr;55(4):1271-81. doi: 10.1002/hep.24792. Epub 2012 Mar 1. PMID 22095555